CLINICAL TRIAL: NCT05962905
Title: Medtronic Accuracy Performance Verification of the INVOS™ System in the Pediatric Cardiac Catheterization Laboratory (INCATH)
Brief Title: Accuracy Performance Verification of the INVOS™ System in Pediatrics
Acronym: INCATH
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT23002INCATH
Record Dates: First submitted 2023-07-13; First posted 2023-07-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Oxygenation; Pediatric ALL
Keywords: cerebral oximetry; pediatric; infant
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pediatric: Subjects meeting inclusion criteria weighing between 4 and 40 kg
  Interventions: Other: Blood sample; Device: INVOS monitoring
- Infant: Subjects meeting inclusion criteria weighing under 40 kg
  Interventions: Other: Blood sample; Device: INVOS monitoring

INTERVENTIONS:
Other: Blood sample — During the standard of care interventional or diagnostic cardiac catheterization, paired arterial and venous blood samples will be obtained. The venous sample will be obtained from 2 cm superior to the clavicle, which is beyond standard of care during the routine cardiac catheterization
Device: INVOS monitoring — During the standard of care interventional or diagnostic cardiac catheterization, INVOS monitoring will be used. INVOS™ regional oxygen saturation (rSO2) values will be compared to the calculated global field saturation of cerebral tissue determined from blood sample co-oximetry.

SUMMARY:
Prospective, observational, multi-center trial designed to capture calibration and performance evaluation data with the INVOS™ system.

DETAILED DESCRIPTION:
The purpose of this study is to verify INVOS™ cerebral oximetry system performance in pediatric and infant patients bycomparing regional oxygen saturation (rSO2) values to reference blood oxygen saturation measurements obtained throughinternal jugular vein and arterial blood convenience sampling according to International Organization on Standards (ISO) 80601-2-85:2021.

ELIGIBILITY:
Inclusion Criteria:

1. Under 21 years of age
2. Meets weight requirement for sensors under study
3. Scheduled for a diagnostic or interventional cardiac catheterization procedure with general anesthesia or sedation
4. Arterial and venous access as part of the planned catheterization procedure

Exclusion Criteria:

1. Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported]
2. A skin condition at the sensor site (e.g., rash, abrasion, laceration)
3. Craniofacial disease producing abnormal forehead anatomy and/or preventing forehead application of the sensor
4. A known structural brain lesion beneath the sensor
5. Known hemoglobinopathy
6. Inability to lie supine with neutral neck position during catheterization
7. Cerebrovascular disease
8. An emergent, life threatening condition impacting study conduct
9. Unwillingness or inability to sign informed consent (IC) or assent by the parents/guardians of child
10. Currently receiving phototherapy for bilirubin
11. Arterial or venous anatomy that would preclude obtaining an accurate paired sample
12. Known pregnancy

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (under 21) weighing under 40 kg scheduled for a diagnostic or interventional cardiac catheterization procedure with general anesthesia or sedation
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the root mean square | At the point of blood sampling during cardiac catheterization procedure
  root mean square of the difference in regional oxygen saturation (rSO2) as measured by the INVOS and field saturation (fSO2) as measured by blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Ami R Stuart, PhD, Study Director — Principal Clinical Research Specialist
Locations (5):
- United States (5):
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No